CLINICAL TRIAL: NCT06441929
Title: How Difficult a Fetal Ultrasound Can be: Time for a Dedicated Classification System
Brief Title: Pregnancy Ultrasound Satisfaction Scoring System
Acronym: 1/2024
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Roberta Zupo, PhD, University of Bari Aldo Moro
Other Study IDs: 1/2024
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Ultrasound Satisfaction in Pregnant Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sonographic imaging stands as the mainstay of fetal anatomical investigation and the primary screening tool for structural abnormalities early in pregnancy. This study aimed to evaluate the occurrence and effect of a cluster of maternal features on sonographic image quality and operator satisfaction.

DETAILED DESCRIPTION:
This was a cross-sectional, single-center observational study of ultrasound scans performed on singleton pregnant women who underwent ultrasound imaging at 11-14 weeks and 19-21 weeks gestation. From March 2023 to March 2024, a convenience cohort of pregnant women who presented for prenatal care at the Fetal Medicine and Prenatal Diagnosis Unit of "Di Venere" Hospital in Bari (Apulia, Southern Italy) and the Obstetrics and Gynecology Unit of Vito Fazzi Hospital in Lecce (Apulia, Southern Italy) to receive routine gestational ultrasound was recruited for the present study.

The inclusion criteria were singleton pregnancy and the presence of one or more of the risk factors widely described in the literature as limiting features, i.e., excess weight (BMI>24.9 Kg/m2), retroverted uterus, the presence of myomas, a previous abdominal surgery, and a limited echo absorption. No exclusion criteria related to women's gestational age or ethnicity were applied.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women presenting one or more of the risk factors widely described in the literature as limiting features, i.e., excess weight (BMI>24.9 Kg/m2), retroverted uterus, the presence of myomas, previous abdominal surgery, and limited echo absorption.

Exclusion Criteria:

* No limiting factors described above
* No pregnant women

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women presenting one or more of the risk factors widely described in the literature as limiting features, i.e., excess weight (BMI>24.9 Kg/m2), retroverted uterus, the presence of myomas, previous abdominal surgery, and limited echo absorption.
Study Population: A cohort of pregnant women who underwent ultrasound imaging at 11-14 weeks and 19-21 weeks gestation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Operator ultrasound satisfaction | baseline
  Operator ultrasound satisfaction, rating as "low", "good", or "very good"

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bari Aldo Moro, Bari, Italy

IPD SHARING:
Plan to Share IPD: No